CLINICAL TRIAL: NCT06957288
Title: The Effect of Mindfulness-Based Death Psychoeducation Program on Death Awareness and Death Anxiety Levels in Nurses
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kastamonu University (Other)
Responsible Party: Principal Investigator, Havva Kaçan, ASSOCIATE PROFESSOR, Kastamonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025/3/41
Record Dates: First submitted 2025-04-26; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Death Anxiety; Death Occurring in Intensive Care Units
Keywords: Death Anxiety; death awareness; Nurse
MeSH Terms: conditions — Necrophobia

STUDY DESIGN:
Intervention Model Description: The study will include nurses working at Kastamonu University Education and Research Hospital. All nurses will be informed about the nature of the interviews and scales, and written informed consent will be obtained from nurses who accept the evaluation. Written permission will be obtained from the Provincial Health Directorate for the study. The study group nurses will be divided into two groups and the training will be given once a week in two forty-five minute lessons in 12 sessions and will be completed in approximately 6 weeks.
  -Research Universe/Sample or Study Group: Nurses working at Kastamonu University Education and Research Hospital will constitute the universe, and nurses who accept to participate in the study will constitute the sample. Power analysis will be conducted to determine the number of people to be included in the sample, and will be calculated with the G*Power 3.1 program. Power analysis will be conducted to determine the number of people to be included .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Awareness-Based Psychoeducation (Experimental): The aim of psychoeducation is to reduce the death anxiety of nurses and to increase their awareness of death by providing them with information about the death experience they are secondarily exposed to (1- Death process and death anxiety, 2- Effects of the death process on the individual and family, 3- Coping with the death process, 4- Effects of the death process on caregiving nurses, 5- Awareness of death, 6- Nursing care and emotional competence during the death process). Therefore, it will be evaluated whether the implemented psychoeducation program reduces the intended death anxiety and creates awareness about death. This study will be conducted to examine the effect of a 6-week, 12-session mindfulness-based group psychoeducation program given to nurses on death anxiety and death awareness levels.
  Interventions: Other: Mindfulness-based psychoeducation

INTERVENTIONS:
Other: Mindfulness-based psychoeducation — The aim of psychoeducation is to reduce the death anxiety of nurses and to increase their awareness of death by providing them with information about the death experience they are secondarily exposed to (1- Death process and death anxiety, 2- Effects of the death process on the individual and family, 3- Coping with the death process, 4- Effects of the death process on caregiving nurses, 5- Awareness of death, 6- Nursing care and emotional competence during the death process). Therefore, it will be evaluated whether the implemented psychoeducation program reduces the intended death anxiety and creates awareness about death. This study will be conducted to examine the effect of a 6-week, 12-session mindfulness-based group psychoeducation program given to nurses on death anxiety and death awareness levels.

SUMMARY:
Nurses are the primary caregivers for individuals who experience difficult situations (disease, loss, etc.) or are in the terminal phase. This may cause nurses to be exposed to the same experiences secondarily. Coming face to face with death can be a traumatic experience for individuals. Whether death is a traumatic experience for nurses may vary depending on individual differences and environmental conditions. Factors affecting nurses in this sense include the unit they work in, death anxiety, death awareness, workload, and sociodemographic characteristics. Studies conducted with nurses indicate that nurses' death anxiety varies depending on the unit and other factors, and that nurses need training for death awareness and the right approach to individuals. A study conducted on death education and grief counseling determined that individuals' participation in death education does not always help them cope with death and grief, but that individuals can be significantly helped in the face of death and loss if individual differences in coping with grief are focused on and helping skills are developed.

It is thought that the awareness-based death-themed psychoeducation program to be applied to nurses in line with their educational needs will increase nurses' death awareness and reduce their death anxiety levels. The nurses working at Kastamonu Education and Research Hospital will constitute the universe of the study. The research will be conducted with nurses in a pre-test-post-test, experimental and control group experimental design. A power analysis will be conducted to determine the number of people to be included in the sample.

It will be calculated with G*Power 3.1 program. In the sample calculation, effect size (d=1.1), 5% margin of error (α=0.05) and power (1-β=0.95) were taken into account and 30 people were needed in the groups, 15 experimental and 15 control. However, considering the data loss, the sample size for each group was increased by 20% and it was planned to include 18 people in each group, a total of 36 people in the sample. In addition to descriptive statistical methods (Mean, Standard deviation) in the evaluation of the data, correlation test will be used to evaluate the relationship between the mean scores before and after the education in the comparison of quantitative data. Wilcoxon Associated Sample Test will be used to make comparisons before and after the education. ''Nurses Descriptive Information Form'', ''Multidimensional Death Awareness Scale'' and ''Thorson Powell Death Anxiety Scale'' will be used in the collection of data. A mindfulness-based psychoeducation program will be applied to the experimental group. The aim of the psychoeducation is to reduce the death anxiety of the nurses and to increase their awareness of death by providing them with information about the death experience they are secondarily exposed to (1- Death process and death anxiety, 2- Effects of the death process on the individual and family, 3- Coping with the death process, 4- Effects of the death process on caregiving nurses, 5- Awareness of death, 6- Nursing care and emotional competence during the death process). Therefore, it will be evaluated whether the applied psychoeducation program reduces the intended death anxiety and creates awareness about death. This study will be conducted to examine the effect of a 6-week, 12-session mindfulness-based group psychoeducation program given to nurses on death anxiety and death awareness levels.

DETAILED DESCRIPTION:
Nurses are the primary caregivers for individuals who experience difficult situations (disease, loss, etc.) or are in the terminal phase. This may cause nurses to be exposed to the same experiences secondarily. Coming face to face with death can be a traumatic experience for individuals. Whether death is a traumatic experience for nurses may vary depending on individual differences and environmental conditions. Factors affecting nurses in this sense include the unit they work in, death anxiety, death awareness, workload, and sociodemographic characteristics. Studies conducted with nurses indicate that nurses' death anxiety varies depending on the unit and other factors, and that nurses need training for death awareness and the right approach to individuals. A study conducted on death education and grief counseling determined that individuals' participation in death education does not always help them cope with death and grief, but that individuals can be significantly helped in the face of death and loss if individual differences in coping with grief are focused on and helping skills are developed.

It is thought that the awareness-based death-themed psychoeducation program to be applied to nurses in line with their educational needs will increase nurses' death awareness and reduce their death anxiety levels. The nurses working at Kastamonu Education and Research Hospital will constitute the universe of the study. The research will be conducted with nurses in a pre-test-post-test, experimental and control group experimental design. A power analysis will be conducted to determine the number of people to be included in the sample.

It will be calculated with G*Power 3.1 program. In the sample calculation, effect size (d=1.1), 5% margin of error (α=0.05) and power (1-β=0.95) were taken into account and 30 people were needed in the groups, 15 experimental and 15 control. However, considering the data loss, the sample size for each group was increased by 20% and it was planned to include 18 people in each group, a total of 36 people in the sample. In addition to descriptive statistical methods (Mean, Standard deviation) in the evaluation of the data, correlation test will be used to evaluate the relationship between the mean scores before and after the education in the comparison of quantitative data. Wilcoxon Associated Sample Test will be used to make comparisons before and after the education. ''Nurses Descriptive Information Form'', ''Multidimensional Death Awareness Scale'' and ''Thorson Powell Death Anxiety Scale'' will be used in the collection of data. A mindfulness-based psychoeducation program will be applied to the experimental group. The aim of the psychoeducation is to reduce the death anxiety of the nurses and to increase their awareness of death by providing them with information about the death experience they are secondarily exposed to (1- Death process and death anxiety, 2- Effects of the death process on the individual and family, 3- Coping with the death process, 4- Effects of the death process on caregiving nurses, 5- Awareness of death, 6- Nursing care and emotional competence during the death process). Therefore, it will be evaluated whether the applied psychoeducation program reduces the intended death anxiety and creates awareness about death. This study will be conducted to examine the effect of a 6-week, 12-session mindfulness-based group psychoeducation program given to nurses on death anxiety and death awareness levels.In this study, the death psychoeducation applied to nurses will provide psychological support to nurses, help nurses manage the anxiety they experience when faced with death and experience low levels of death anxiety, and will also support the acceptance of death as a reality and the increase in their awareness of death. It is thought that with the increased awareness of death, nurses who are primary caregivers will also make positive contributions to nursing care.

ELIGIBILITY:
Inclusion Criteria:

* Working as a nurse in Palliative Care services, emergency services and intensive care units

Exclusion Criteria:

* Working as a nurse outside of Palliative Care services, emergency services and intensive care units

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-10 (Estimated); Primary Completion 2025-06-10 (Estimated); Study Completion 2025-07-10 (Estimated)

PRIMARY OUTCOMES:
The death anxiety level of nurses who participate in psychoeducation will decrease. | Four Week
  The death anxiety level of nurses participating in psychoeducation will be measured with the Thorson Powell death anxiety scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Kastamonu Hospital, Kastamonu, Central, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
ı don't want